CLINICAL TRIAL: NCT04258059
Title: Wells and Enteric Disease Transmission - A Randomized Controlled Trial (WET- Trial)
Brief Title: Wells and Enteric Disease Transmission Trial (WET - Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Principal Investigator, Heather Murphy, Adjunct Associate Research Professor, Temple University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 25665 (Pilot Trial)
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Infection; Respiratory Viral Infection
Keywords: groundwater; private wells; acute gastrointestinal illness; respiratory infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active UV Device (Active Comparator): A household water treatment device with a lamp emitting germicidal UV. The device will be operated at 50 millijoule per square centimeter to treat >99.9% of all bacteria, protozoa, and most viruses in water supplies.
  Interventions: Device: Active household UV water treatment device
- Inactive UV Device (Sham Comparator): A device that appears identical to the active comparator device except the lamp will not emit germicidal UV.
  Interventions: Device: Inactive household UV water treatment device

INTERVENTIONS:
Device: Active household UV water treatment device — This point-of-entry treatment device will use germicidal UV to treat all of the well water used in the home.
  Arms: Active UV Device
Device: Inactive household UV water treatment device — This sham device will use a lamp not emitting germicidal UV.
  Arms: Inactive UV Device

SUMMARY:
Approximately 40 million people in the US are served by private wells, many of which are untreated. The investigators estimate that 1.29 million cases of gastrointestinal illness (GI) per year are attributed to consuming water from untreated private wells in the US. These cases of GI can cause a significant burden in terms of health care costs and lost work/school days, as well as increased risk to developing longer term health complications. This impact is magnified when accounting for vulnerable populations such as children under the age of 5, the elderly and the immunocompromised. The investigators are preparing to conduct the first household randomized controlled trial (RCT) to investigate whether consuming well water treated by ultraviolet light (UV) compared to consuming untreated private well water decreases the incidence of self-reported gastrointestinal illness and respiratory infections in children under 5. The investigators will collect illness symptom data using a combination of weekly text messages and online illness questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Child resides in Berks, Bucks, Chester, Lancaster, Lehigh, or Montgomery County in Pennsylvania
* Household is served by a private well
* Participant child is under the age of 5 (under 4 at time of enrollment), who is a full-time resident of the home and drinks untreated well water (75% or more of water consumption must be from untreated well water)
* Parent/guardian has access to a phone with texting capabilities

Exclusion Criteria:

* Child participant is immunocompromised
* Child participant has a chronic gastrointestinal condition
* Child takes daily oral steroids
* Household treats water before consumption (with the exception of water softeners)

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Incident gastrointestinal illness | 12 months
  The investigators will collect data on the presence of gastrointestinal illness symptoms through weekly text messages. Households that report symptoms through text messages will be directed to an online illness questionnaire to characterize the symptoms (incidence, severity, duration, diarrhea, vomiting, coughing, etc.), febrile episodes, as well as relevant exposure information such as recent travel, exposure to ill persons, etc. Incident gastrointestinal illness (GI) is defined by the reporting of a minimum of three episodes of diarrhea or vomiting in a 24 hour period. Each illness will be considered distinct when separated by ≥ 6 symptom-free days.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Murphy, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hellard ME, Sinclair MI, Harris AH, Kirk M, Fairley CK. Cost of community gastroenteritis. J Gastroenterol Hepatol. 2003 Mar;18(3):322-8. doi: 10.1046/j.1440-1746.2003.02959.x. PMID 12603534
- [Background] Johnson TD, Belitz K, Lombard MA. Estimating domestic well locations and populations served in the contiguous U.S. for years 2000 and 2010. Sci Total Environ. 2019 Oct 15;687:1261-1273. doi: 10.1016/j.scitotenv.2019.06.036. Epub 2019 Jun 6. PMID 31412460
- [Background] Roberts JA, Cumberland P, Sockett PN, Wheeler J, Rodrigues LC, Sethi D, Roderick PJ; Infectious Intestinal Disease Study Executive. The study of infectious intestinal disease in England: socio-economic impact. Epidemiol Infect. 2003 Feb;130(1):1-11. doi: 10.1017/s0950268802007690. PMID 12613740